CLINICAL TRIAL: NCT00893100
Title: Evaluation of Pain Reduction After Hemorrhoidectomy With Use of Diltiazim Ointment 2%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Bagher Larijani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 724
Record Dates: First submitted 2009-04-19; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diltiazem (Experimental)
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Diltiazem — 2%,3 times daily

SUMMARY:
The purpose of this study is to evaluate the effectiveness of diltiazem ointment 2 percent in reducing pain after hemorrhoidectomy.

DETAILED DESCRIPTION:
Pain after hemorrhoidectomy remains a major postsurgical complication.Therefore pain management in patients is an important goal.Many studies have focused on surgical techniques,preoperative and postoperative regimes.We assessed a randomised double blind placebo-controlled trial to evaluate the effect of diltiazem ointment after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade 3 or 4 hemorrhoid who underwent Milligan-Morgan surgery.

Exclusion Criteria:

* Patients with a history of heart disease, blood pressure, orthostatic hypertension, hemorrhoidal surgery,or those who had previous adverse effect from calcium channel blocker drugs and also those who were pregnant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Reduction of Pain | daily in one week

CONTACTS AND LOCATIONS:
Overall Officials: Farshad Jalili, Resident, Principal Investigator — Sina Hospital
Locations (1):
- Sina General Hospital, Tehran, Tehran Province, Iran